CLINICAL TRIAL: NCT02766400
Title: Guided Versus Directed Training in Acute Stroke Rehabilitation
Brief Title: Examining Rehabilitation Training Methods
Acronym: GUIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Elizabeth R. Skidmore, PhD, OTR/L, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO12040383; R03HD073770-01 (NIH); R01HD074693-02S1 (NIH); UL1TR000005 (NIH)
Record Dates: First submitted 2016-05-03; First posted 2016-05-09 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Guided Training; Directed Training
Keywords: Stroke; Rehabilitation; Cognition; Disability; Intervention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guided Training (Experimental): Guided training is a rehabilitation training approach that maximizes the expertise of the patient, by teaching patients to identify and prioritize activities, identify barriers to performing activities, generate their own strategies for addressing these barriers, and apply this process through iterative practice. Guided training equips patients with "practical" skills that have the potential to generalize beyond activities addressed during the intervention program to novel problematic activities that arise after the intervention program, thereby promoting long-term independence.
  Interventions: Behavioral: Guided Training
- Directed Training (Active Comparator): Directed training is a rehabilitation approach that maximizes the expertise of the rehabilitation practitioner. Rehabilitation practitioners identify and prioritize problematic activities, identify barriers to performing these activities, generate strategies to address these barriers and instruct patients in these strategies, and repeat the process with a variety of problematic activities identified during the rehabilitation program. Directed training promotes independence with training activities, however the benefits of direct training are likely to be activity-specific (i.e., only promote improvement on the trained activity) and not generalizable to other daily activities. This therapist-directed approach is currently the method used most frequently in acute rehabilitation.
  Interventions: Behavioral: Directed Training

INTERVENTIONS:
Behavioral: Guided Training
  Other Names: Strategy Training
  Arms: Guided Training
Behavioral: Directed Training
  Other Names: Direct Skill Training
  Arms: Directed Training

SUMMARY:
Individuals with cognitive impairments after stroke sustain significant disability in their daily tasks, and account for a significant proportion of stroke-related healthcare costs. This loss of independence is costly because individuals with stroke-related cognitive impairments require more rehabilitation and more resources to support their living, whether in institutional or community settings. The proposed study examines the effects of directed and guided training on the recovery of independence with daily activities in adults with stroke-related cognitive impairments in acute rehabilitation. The investigators predict that patients in both groups will demonstrate significant improvement in independence with daily activities in the first 12 months after rehabilitation admission, but that patients who receive guided training will demonstrate significantly more improvements than patients who received directed training.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of acute stroke
* admission to acute inpatient rehabilitation
* impairment in cognitive functions (as indicated by 14-item Executive Interview ≥ 3)

Exclusion Criteria:

* diagnosis of dementia in the medical record
* inability to follow two-step commands 80% of the time
* severe aphasia (score of 0 or 1 on the Boston Diagnostic Aphasia Examination 3rd Edition Severity Rating Scale)
* current untreated major depressive, bipolar, or psychotic disorder (PRIME-MD)
* drug or alcohol abuse within 3 months (Mini-International Neuropsychiatric Interview)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Skidmore, PhD, OTR/L, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
At present, there is no plan to share data.

REFERENCES:
- [Derived] Kringle EA, Terhorst L, Butters MA, Skidmore ER. Clinical Predictors of Engagement in Inpatient Rehabilitation Among Stroke Survivors With Cognitive Deficits: An Exploratory Study. J Int Neuropsychol Soc. 2018 Jul;24(6):572-583. doi: 10.1017/S1355617718000085. Epub 2018 Mar 19. PMID 29552996
- [Derived] Skidmore ER, Butters M, Whyte E, Grattan E, Shen J, Terhorst L. Guided Training Relative to Direct Skill Training for Individuals With Cognitive Impairments After Stroke: A Pilot Randomized Trial. Arch Phys Med Rehabil. 2017 Apr;98(4):673-680. doi: 10.1016/j.apmr.2016.10.004. Epub 2016 Oct 26. PMID 27794487

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: August 2012 to December 2014. Participants with acute stroke were enrolled in inpatient rehabilitation at Mercy and Montefiore Hospital.
Pre-assignment Details: Excluded (n=27)
  * Insufficient cognitive impairment (n=6)
  * Mood/psychotic disorder (n=14)
  * Drug/alcohol abuse (n=3)
  * Change in medical status (n=1)
  * Pre-morbid cognitive impairment (n=1)
  * Short Length of Stay (n=2)
  Withdrew prior to randomization (n=7)
  * Changed mind (n=4)
  * Discharged (n=3)
Groups:
- Guided Training: Guided training is a rehabilitation training approach that maximizes the expertise of the patient, by teaching patients to identify and prioritize activities, identify barriers to performing activities, generate their own strategies for addressing these barriers, and apply this process through iterative practice. Guided training equips patients with "practical" skills that have the potential to generalize beyond activities addressed during the intervention program to novel problematic activities that arise after the intervention program, thereby promoting long-term independence.
  Guided Training
- Directed Training: Directed training is a rehabilitation approach that maximizes the expertise of the rehabilitation practitioner. Rehabilitation practitioners identify and prioritize problematic activities, identify barriers to performing these activities, generate strategies to address these barriers and instruct patients in these strategies, and repeat the process with a variety of problematic activities identified during the rehabilitation program. Directed training promotes independence with training activities, however the benefits of direct training are likely to be activity-specific (i.e., only promote improvement on the trained activity) and not generalizable to other daily activities. This therapist-directed approach is currently the method used most frequently in acute rehabilitation.
  Directed Training
Period: Overall Study
Arm/Group | Guided Training | Directed Training
Started | 21 | 22
Completed | 19 | 20
Not Completed | 2 | 2
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guided Training | Directed Training | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.86 (11.67) | 66.73 (14.25) | 66.30 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 9 | 13 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20 | 21 | 41
  African American | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 43
Stroke onset [Mean (Standard Deviation); unit: days] — Stroke onset is calculated from date of stroke to date of study admission.
  days | 16.29 (18.24) | 22.36 (30.97) | 19.40 (25.46)
Stroke type [Number; unit: participants]
  ischemic | 14 | 14 | 28
  hemorrhagic | 7 | 8 | 15
Hemisphere [Number; unit: participants]
  Left | 10 | 13 | 23
  Right | 11 | 9 | 20
Stroke severity, NIHSS [Mean (Standard Deviation); unit: units on a scale] — The NIHSS is composed of 11 items that are summed to yield a total score. Total scores range from 0 to 42, where 0=no neurological impairment, and 42=severe neurological impairment.
  units on a scale | 7.00 (3.90) | 7.86 (5.10) | 7.44 (4.52)
Cognitive status, EXIT [Mean (Standard Deviation); unit: units on a scale] — The EXIT is composed of 14 items that are summed to yield a total score ranging from 0 to 28. A total score of 0 typically indicates no executive impairment, while a total score of 28 indicates severe executive impairment.
  units on a scale | 12.38 (5.11) | 10.86 (5.14) | 11.60 (5.12)
Functional Independence Measure [Mean (Standard Deviation); unit: units on a scale] — The Functional Independence Measure contains 18 items composed of 13 motor tasks and 5 cognitive tasks. A total score of 18-126 is obtained where 18 represents complete dependence/total assistance and 126 represents complete independence with daily activities.
  units on a scale | 67.33 (14.72) | 67.32 (18.33) | 67.33 (16.47)

OUTCOME MEASURES:

1. Primary Outcome: Differences in Independence With Activities of Daily Living (Functional Independence Measure) Between Groups Over Time
Description: Differences between groups in mean independence scores (computed from Functional Independence Measure total scores) over time.
  The Functional Independence Measure contains 18 items with a total score ranging from 18-126 is obtained (18=complete dependence/total assistance with basic self-care and mobility activities; 126=complete independence with basic self-care and mobility activities). Total scores were calculated for each participant at baseline, discharge, month 3, month 6, and month 12, and mean total scores for each group were calculated at each time point. Differences in mean scores were examined between groups over time with mixed model analyses.
Time Frame: Baseline, rehab discharge, month 3, month 6, month 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Guided Training | Directed Training
Number analyzed (Participants) | 21 | 22
units on a scale
  Baseline Scores | 67.33 (3.21) | 67.32 (3.91)
  Discharge Scores | 86.86 (3.08) | 89.05 (4.41)
  Month 3 Scores | 105.32 (4.94) | 102.55 (5.41)
  Month 6 Scores | 107.68 (3.45) | 100.52 (5.35)
  Month 12 Scores | 108.47 (4.34) | 100.25 (5.12)
Statistical Analysis 1: Comparison: Guided Training vs Directed Training; All analyses were performed using the intent-to-treat principle so that comparisons were made according to the assigned intervention group regardless of study completion; Test type: Superiority or Other; p < 0.001, Linear mixed models — a priori threshold was set at p<0.05; F(4,150)=5.11; Cohen's d effect size at 12 months = 0.53, 95% CI 2-sided [-0.12 to 1.19] — Effect size was calculated using mean change scores (baseline to month 12) and standard error of change (baseline to month 12) for each group

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Guided Training | Directed Training
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22

LIMITATIONS AND CAVEATS:
Both interventions were offered in addition to usual care (comprised mostly of direct skill training). This may have minimized the overall effect of guided training.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes